CLINICAL TRIAL: NCT01909375
Title: American Joint Replacement Registry
Acronym: AJRR
Status: Recruiting | Type: Observational
Sponsor: American Joint Replacement Registry (Other)
Responsible Party: Principal Investigator, Nathan Glusenkamp, Chief Quality and Registries Officer, American Joint Replacement Registry
Other Study IDs: 1120353
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: ARTHROPLASTY, REPLACEMENT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The American Joint Replacement Registry is a not-for-profit 501(c)(3) organization for data collection and quality improvement initiatives for total hip and knee replacements. The AJRR is a collaborative effort supported by the American Academy of Orthopaedic Surgeons (AAOS), the American Association of Hip and Knee Surgeons (AAHKS), The Hip Society, The Knee Society, hospitals, health insurers, medical device manufacturers, and contributions from individual orthopaedic surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Any individual in the US undergoing total joint arthroplasty

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We expect to receive data on up to 90% of all total joint arthroplasties conducted in the United States annually.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | 12 months
  Utilization of VR-12 and/or PROMIS-10

SECONDARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score - Joint Replacement (HOOS, JR) | 12 months

OTHER OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - Joint Replacement (KOOS, JR) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Glusenkamp, Principal Investigator — American Joint Replacement Registry; David G Lewallen, MD, Study Director — American Joint Replacement Registry
Locations (1):
- Nathan Glusenkamp, Rosemont, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
AJRR provides participating hospitals their data back in the form of dashboards and reports available on our registry platform. AJRR also releases an Annual Report every November which includes aggregate, de-identified data.